CLINICAL TRIAL: NCT00578981
Title: Wiser Choices in Osteoporosis Trial: The OSTEOPOROSIS CHOICE Decision Aid to Support the Decision to Use or Not Use Bisphosphonates in Postmenopausal Women at Risk of Osteoporotic Fractures.
Brief Title: Osteoporosis Choice Decision Aid for Use of Bisphosphonates in Postmenopausal Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Victor Montori, MD, Mayo Clinic
Allocation: Randomized | Model: Factorial | Masking: Single
Other Study IDs: 07-003475
Record Dates: First submitted 2007-12-20; First posted 2007-12-21 (Estimated); Last update posted 2016-02-02 (Estimated); Status verified 2016-02

CONDITIONS: Osteoporosis; Bone Loss, Age Related; Postmenopausal Bone Loss; Postmenopausal Osteoporosis
Keywords: Osteoporosis, age-related; Osteoporosis, Postmenopausal; Bone Loss; Low Bone Density
MeSH Terms: conditions — Osteoporosis; Osteoporosis, Postmenopausal; Bone Diseases, Metabolic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Behavioral: Osteoporosis Choice Decision Aid
- Arm 2 (No Intervention)

INTERVENTIONS:
Behavioral: Osteoporosis Choice Decision Aid — The provider will introduce the patient to the choice of bisphosphonates using the decision aid.
  Arms: Arm 1

SUMMARY:
To develop a decision aid to support the decision to use (or not use) bisphosphonates in postmenopausal women at risk for osteoporotic fractures, and to assess the impact of the decision aid on start and six month adherence to bisphosphonates.

DETAILED DESCRIPTION:
Bisphosphonates can reduce fracture risk in patients with osteoporosis. However, many patients may not start and adhere to bisphosphonates, consequently losing independence, quality, and length of life. We hypothesize that a decision aid that efficiently improves patient education and communication with their provider about fracture risk, and about using bisphosphonates to reduce that risk, will improve the quality of treatment decisions. We anticipate that patients will become more involved in the decision-making process and decisions will be more consistent with patients' values and health care goals. We expect this will lead to increased bisphosphonate start and adherence and improved patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Female, post-menopausal women aged 50 to 90.
* Have a bone mineral density (BMD) evaluation resulting in a T-Score of <-1.0.
* Have a follow-up appointment with a provider in the areas of Family Medicine (FM), Primary Care Internal Medicine (PCIM), or POM.
* Have no major barriers (i.e., severe hearing impairment, dementia, require interpreter, etc.) to participation in shared decision-making (per provider's assessment)
* Enrollment is open to females of diverse racial backgrounds.

Exclusion Criteria:

* Currently taking a bisphosphonate.
* Not available for 6 month follow-up phone call.

Ages: 50 Years to 90 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2007-08; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Evidence of success of decision aid to providers and patients, which leads to improved knowledge, reduced decisional conflict and enhanced satisfaction with the decision, and enhanced adherence to medication. | Directly following intervention.

SECONDARY OUTCOMES:
Evaluate ability to recruit participants and collect patient outcomes. | One year after start of study.

CONTACTS AND LOCATIONS:
Overall Officials: Victor M. Montori, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Wyatt KD, Branda ME, Inselman JW, Ting HH, Hess EP, Montori VM, LeBlanc A. Genders of patients and clinicians and their effect on shared decision making: a participant-level meta-analysis. BMC Med Inform Decis Mak. 2014 Sep 2;14:81. doi: 10.1186/1472-6947-14-81. PMID 25179289
- [Derived] Montori VM, Shah ND, Pencille LJ, Branda ME, Van Houten HK, Swiglo BA, Kesman RL, Tulledge-Scheitel SM, Jaeger TM, Johnson RE, Bartel GA, Melton LJ 3rd, Wermers RA. Use of a decision aid to improve treatment decisions in osteoporosis: the osteoporosis choice randomized trial. Am J Med. 2011 Jun;124(6):549-56. doi: 10.1016/j.amjmed.2011.01.013. PMID 21605732
- [Derived] Pencille LJ, Campbell ME, Van Houten HK, Shah ND, Mullan RJ, Swiglo BA, Breslin M, Kesman RL, Tulledge-Scheitel SM, Jaeger TM, Johnson RE, Bartel GA, Wermers RA, Melton LJ 3rd, Montori VM. Protocol for the Osteoporosis Choice trial. A pilot randomized trial of a decision aid in primary care practice. Trials. 2009 Dec 10;10:113. doi: 10.1186/1745-6215-10-113. PMID 20003299